CLINICAL TRIAL: NCT00607737
Title: Doubleblind, Randomised, Single Centre Investigator Sponsored Study of Applications Site Reactions After Deep and Superficial Subcutaneous and Intradermal Injection of Insulin Detemir and Saline in Subjects With Diabetes Mellitus
Brief Title: Applications Site Reactions After Injection of Insulin Detemir and Saline in Subjects With Diabetes
Acronym: APPLY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lise Tarnow (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor-Investigator, Lise Tarnow, professor, Steno Diabetes Center Copenhagen
Organization: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: APPLY; EudraCT 2007-005677-59
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Detemir; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): insulin detemir
  Interventions: Drug: insulin detemir
- 2 (Placebo Comparator): saline
  Interventions: Drug: saline

INTERVENTIONS:
Drug: insulin detemir — 3 cutaneous injections
  Arms: 1
Drug: saline — 3 cutaneous injections
  Arms: 2

SUMMARY:
To compare application site reactions after superficial and deep subcutaneous and intradermal injections of insulin detemir and saline in patients with diabetes

- The patient serves as his own control, n=100 patients with diabetes

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus
* HbA1c<11 %
* BMI: 20-35 kg/m2
* Insulin detemir naive
* Basal insulin dose>20E

Exclusion Criteria:

* Known allergy to study drug
* Current steroid or antiallergic treatment
* Lipodystrophy
* Change in insulin and antihypertensive treatment < 30 days
* Smokers or alcoholics

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
laser doppler blood flow | 10 minutes - 7 days

SECONDARY OUTCOMES:
clinical signs | 10 min - 7 days
insulin detemir specific antibodies | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: LIse Tarnow, md, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Denmark

REFERENCES:
- See also: publication — http://onlinelibrary.wiley.com/doi/10.1111/j.1600-0846.2011.00551.x/pdf